CLINICAL TRIAL: NCT01743820
Title: Phase 2a Dose Escalation Study of the Efficacy, Safety, and Pharmacokinetics of Low Dose Primaquine for Gametocytocidal Activity Against P. Falciparum in Sub-Saharan Africa and South East Asia
Brief Title: Phase2a Primaquine Dose Escalation Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Shoklo Malaria Research Unit (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Bill and Melinda Gates Foundation (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEG001; NCT02011555 (obsolete NCT alias)
Record Dates: First submitted 2012-11-26; First posted 2012-12-06 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- dihydroartemisinin-piperaquine only (Active Comparator): dihydroartemisinin -piperaquine (DP) only
  Interventions: Drug: dihydroartemisinin-piperaquine
- DP and 0.125 mg/kg primaquine (Experimental): DP and single dose oral 0.125 mg/kg primaquine
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: 0.125 mg/kg Primaquine
- DP and 0.5 mg/kg primaquine (Experimental): DP and single dose oral 0.5 mg/kg primaquine
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: 0.5 mg/kg Primaquine
- DP and 0.25 mg/kg primaquine (Experimental): DP and a single dose oral 0.25 mg/kg primaquine
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: 0.25 mg/kg Primaquine
- DP and 0.0625 mg/kg primaquine (Experimental): DP and a single dose oral 0.0625 mg/kg primaquine
  Interventions: Drug: dihydroartemisinin-piperaquine; Drug: 0.0625 mg/kg Primaquine

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine
Drug: 0.125 mg/kg Primaquine
  Arms: DP and 0.125 mg/kg primaquine
Drug: 0.5 mg/kg Primaquine
  Arms: DP and 0.5 mg/kg primaquine
Drug: 0.25 mg/kg Primaquine
  Arms: DP and 0.25 mg/kg primaquine
Drug: 0.0625 mg/kg Primaquine
  Arms: DP and 0.0625 mg/kg primaquine

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of low single-dose primaquine for gametocidal activity against P.falciparum among adult glucose-6-phosphate dehydrogenase (G6PD)-normal malaria patients.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age >= 18 years and < 50 years
* Malaria blood thick film positive
* Presence of gametocytes on thick blood film
* Agrees to admission to study ward for 26 hours post diagnosis and available for follow up visits
* No allergies to study drugs
* Hemoglobin >= 8 g/dl
* No evidence of severe or chronic disease
* Written, informed consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
mosquito infectivity assessed through membrane feeding | 7 days
  Baseline, Days 1, 2, 7

SECONDARY OUTCOMES:
gametocyte prevalence and density | 28 days
  Baseline, Hours 2, 6, 12, 24, Days 2, 3, 7, 14, 28
primaquine pharmacokinetics - area under the curve (AUC) of parent drug and metabolite | 24 hours
  Hours 1, 2, 3, 4, 6, 8, 12, 24
asexual parasite prevalence and density | 28 days
  Baseline, Hours 2, 6, 12, 24, Days 2, 3, 7, 14, 28
safety measurements including hemoglobin and signs of hemolysis | 28 days
  Baseline, Days 1, 2, 3, 7, 14, 28

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gosling, MD, PhD, Principal Investigator — University of California, San Francisco; Alassane Dicko, MD, Principal Investigator — Malaria Research and Training Centre; François Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

REFERENCES:
- [Background] Gosling RD, Okell L, Mosha J, Chandramohan D. The role of antimalarial treatment in the elimination of malaria. Clin Microbiol Infect. 2011 Nov;17(11):1617-23. doi: 10.1111/j.1469-0691.2011.03660.x. Epub 2011 Sep 26. PMID 21951597
- [Background] Baird JK, Schwartz E, Hoffman SL. Prevention and treatment of vivax malaria. Curr Infect Dis Rep. 2007 Jan;9(1):39-46. doi: 10.1007/s11908-007-0021-4. PMID 17254503
- [Background] WHO (2011) World Malaria Report 2011. Geneva: World Health Organization.
- [Background] WHO (2010) Guidelines for the treatment of malaria, Second edition. Geneva: World Health Organization
- [Background] El-Sayed B, El-Zaki SE, Babiker H, Gadalla N, Ageep T, Mansour F, Baraka O, Milligan P, Babiker A. A randomized open-label trial of artesunate- sulfadoxine-pyrimethamine with or without primaquine for elimination of sub-microscopic P. falciparum parasitaemia and gametocyte carriage in eastern Sudan. PLoS One. 2007 Dec 12;2(12):e1311. doi: 10.1371/journal.pone.0001311. PMID 18074034
- [Background] Shekalaghe SA, ter Braak R, Daou M, Kavishe R, van den Bijllaardt W, van den Bosch S, Koenderink JB, Luty AJ, Whitty CJ, Drakeley C, Sauerwein RW, Bousema T. In Tanzania, hemolysis after a single dose of primaquine coadministered with an artemisinin is not restricted to glucose-6-phosphate dehydrogenase-deficient (G6PD A-) individuals. Antimicrob Agents Chemother. 2010 May;54(5):1762-8. doi: 10.1128/AAC.01135-09. Epub 2010 Mar 1. PMID 20194698
- [Derived] Dicko A, Brown JM, Diawara H, Baber I, Mahamar A, Soumare HM, Sanogo K, Koita F, Keita S, Traore SF, Chen I, Poirot E, Hwang J, McCulloch C, Lanke K, Pett H, Niemi M, Nosten F, Bousema T, Gosling R. Primaquine to reduce transmission of Plasmodium falciparum malaria in Mali: a single-blind, dose-ranging, adaptive randomised phase 2 trial. Lancet Infect Dis. 2016 Jun;16(6):674-684. doi: 10.1016/S1473-3099(15)00479-X. Epub 2016 Feb 20. PMID 26906747